CLINICAL TRIAL: NCT06816186
Title: Department of Nurse-Midwifery and Women Health Graduate Institute of Nurse Midwifery
Brief Title: The Impact of Multimedia Childbirth Prediction on Parturients and Their Spouses
Acronym: multimedia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 24MMHIS256e
Record Dates: First submitted 2024-12-25; First posted 2025-02-10 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-02

CONDITIONS: Multimedia
Keywords: birth signs, anxiety, self-confidence, number of home visits
MeSH Terms: conditions — Anxiety Disorders | interventions — Multimedia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multimedia (Experimental): When mothers and their spouses reported to the health classroom on the 37-week prenatal check-up day, while the experimental group will receive general care and multimedia birth control education intervention
  Interventions: Behavioral: multimedia
- usual care (Placebo Comparator): usual care
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: multimedia — When mothers and their spouses reported to the health classroom on the 37-week prenatal check-up day, the researcher explained the motivation and process of the research. After the women and their spouses agreed to join the study, they were randomly assigned to the experimental group and the control group. The control group will be given general care guidance, while the experimental group will receive general care and multimedia birth control education intervention, and the mothers and their spouses will download and watch the video through Line, an instant messaging software on their mobile phones.
  Arms: Multimedia
Behavioral: Usual Care — When mothers and their spouses reported to the health classroom on the 37-week prenatal check-up day, The control group will be given general care guidance,
  Arms: usual care

SUMMARY:
Multimedia birth prediction intervention helps mothers and their spouses reduce the number of trips to the hospital, reduce anxiety, and increase self-confidence. A total of 83 couples were accepted for cases, with a 10% attrition rate. so, A total of 95 couples were admitted and divided into the experimental group and the intervention measures were implemented Experimental group. Fill out basic demographic and obstetric variables, self-confidence visual analog scale, situational-trait anxiety scale-situational anxiety part at 37 weeks of pregnancy, at the first visit to the hospital, and one hour after admission to the hospital for delivery

DETAILED DESCRIPTION:
More than 90% of pregnant women are prone to anxiety and fear due to unexpected and uncontrollable birth signs before delivery and because they cannot control their own condition.

Pregnant women who receive prenatal education can reduce their fear, depression, anxiety and stress about childbirth, increase their self-confidence during childbirth, and thus gain a positive childbirth experience. As a quasi-experimental study, cases were accepted using a random method. The number of cases admitted was 83 couples, with a 10% attrition rate. Therefore, a total of 95 couples were admitted and divided into an experimental group and a control group. The experimental group received intervention measures, and the control group received intervention measures.

At 37 weeks of pregnancy, at the first visit to the hospital for examination, and one hour after admission, basic demographic and obstetric variables, self-confidence visual analogy scale, and situational-trait anxiety scale-situational anxiety were filled in, and statistical analysis was performed. The methods were descriptive statistics, independent t test, chi-square test, analysis of variance, generalized estimating equations, and linear regression between the experimental and control groups.

ELIGIBILITY:
1. Low-risk first-time mothers over 20 years old and their spouses
2. Pregnancy >37 weeks, pregnancy <40 weeks
3. Single birth, head position
4. Vaginal producers
5. Those who can listen, speak, read and write Chinese

4. Diagnosed by a doctor as prenatal mental illness 5. The fetus' condition requires admission to a moderate or severe ward or intensive care unit.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2024-02-03 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Self-Confidence Visual Analog Scale | Time range: 37 weeks of pregnancy, first visit to the hospital for examination, one hour of hospitalization
  0 points represent the lowest self-confidence and 10 points represent the highest self-confidence
Situational-Trait Anxiety Inventory-Situational Anxiety Section | Time range: 37 weeks of pregnancy, first visit to the hospital for examination, one hour of hospitalization
  The range is from "1" for almost never to "4" for almost always, with higher total scores indicating a higher level of anxiety in the individual.

CONTACTS AND LOCATIONS:
Locations (1):
- Mackay Memorial Hospital, Hsinchu, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: No